CLINICAL TRIAL: NCT06008262
Title: The Effect of Cold Application on Nausea and Vomiting After Laparoscopic Cholecystectomy
Brief Title: Cold Application Effects on Nausea and Vomiting After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Neslihan Ilkaz, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-81477236-604.01.01-1666
Record Dates: First submitted 2023-08-15; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Nausea and Vomiting
Keywords: Laparoscopic cholecystectomy; Postoperative Nausea and Vomiting; Cold application
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Application Group (Experimental): An ice pack will be applied to the posterior upper neck regions of patients with nausea in Group-I, with an interval of 5 minutes. The vital signs of the patients will be recorded. The severity of nausea and pain of the patients will be evaluated with a numerical rating scale. The effectiveness of its application as perceived by the patient will be evaluated.
  Interventions: Other: Cold Application
- Control Group (No Intervention): In the control group, the severity of nausea and pain will be determined by using a numerical evaluation scale in patients with postoperative nausea. Vital signs will be recorded at this stage. Normal procedures will be applied to these patients within the scope of nursing practices.

INTERVENTIONS:
Other: Cold Application — An ice pack will be applied to the posterior upper neck regions of patients with nausea in Group-I, with an interval of 5 minutes. The vital signs of the patients will be recorded. The severity of nausea and pain of the patients will be evaluated with a numerical rating scale. The effectiveness of its application as perceived by the patient will be evaluated.
  Arms: Cold Application Group

SUMMARY:
This clinical trial aims to test the effect of cold application on postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Nausea and vomiting seen within the first 24 hours after surgery are defined as "Post-Operative Nausea and Vomiting (POBK). Postoperative nausea and vomiting are one of the most common complications of anesthesia. It has been reported that the risk of nausea and vomiting is particularly high after laparoscopic cholecystectomy. It is stated that vagal stimulation and pneumoperitoneum process may trigger this situation in laparoscopic surgeries. Nausea and vomiting after surgery is a very uncomfortable situation for the patient. There are several pharmacological methods to prevent and treat POBK. However, it is stated that the non-pharmacological approach should also be brought to the fore. It is stated that cold reduces molecular activity and causes vasoconstriction. It is stated that cold can slow down the blood flow to the vomiting center in the medulla oblongata and the progression of nausea and vomiting can be slowed down. In this way, it is thought that it will contribute to increasing patient satisfaction and providing cost-effective care.

The study will conduct as a prospective randomized controlled trial. After obtaining verbal and written consent from the patients before and after the surgery, the study will conduct with various data collection forms.

These forms are; the patient data collection form, numerical evaluation scale, preoperative Apfel risk score evaluation form, postoperative nausea severity evaluation form, and perceived effectiveness of the ice pack forms will use. Laparoscopic cholecystectomy will perform and all cases meeting the inclusion criteria will evaluate. Patients will randomize. The ice pack will apply in group-I (n=27), and group II (n=27) will be the control group. An ice pack will be applied to the posterior upper neck regions of patients with nausea in Group-I, at an interval of 5 minutes. The vital signs of the patients will be recorded. The severity of nausea and pain of the patients will be evaluated with a numerical rating scale. The effectiveness of its application as perceived by the patient will be evaluated.

In the control group, the severity of nausea and pain will be determined by using a numerical evaluation scale in patients with postoperative nausea. Vital signs will be recorded at this stage. Standard procedures will be applied to these patients within the scope of nursing practices.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in ASA (American Society of Anesthesiologists) I-II-III class
* Being over 18 years old
* Having received general anesthesia
* Preoperative pain value of 6 or less

Exclusion Criteria:

* Severe nausea in the preoperative period
* Being hypothermic in the postoperative period
* Having had head and neck surgery
* Taking prophylactic antiemetics
* Postoperative pain value of 7 and above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from postoperative nausea degree in a 15 minutes | Within 15 minutes of first sense of postoperative nausea
  In this section, the degree of postoperative nausea will decrease or disappear. This status will evaluate with Numerical Evaluation Scale.
Change from postoperative vomiting in a 15 minutes | Within 15 minutes of first sense of postoperative nausea
  In this section, postoperative vomiting will not occur. This status will evaluate with yes/no question.
Evaluation of cold application effectiveness | Within 15 minutes of first sense of postoperative nausea
  In this section, the effectiveness of cold application with a Ice Pack Perceived Effectiveness Form. In this form, there are three different expressions as the application reduced nausea, did not affect nausea, increased nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Ilkaz, PhD, Principal Investigator — Ankara Medipol University
Locations (1):
- Neslihan Ilkaz, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Son JS, Oh JY, Ko S. Effects of hypercapnia on postoperative nausea and vomiting after laparoscopic surgery: a double-blind randomized controlled study. Surg Endosc. 2017 Nov;31(11):4576-4582. doi: 10.1007/s00464-017-5519-8. Epub 2017 Apr 7. PMID 28389799
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Hooper VD. SAMBA Consensus Guidelines for the Management of Postoperative Nausea and Vomiting: An Executive Summary for Perianesthesia Nurses. J Perianesth Nurs. 2015 Oct;30(5):377-82. doi: 10.1016/j.jopan.2015.08.009. No abstract available. PMID 26408511
- [Background] Scharfenberg DR, Salcido A, Malone P, Clark J, Steele MA. Managing Postoperative Nausea With an Application of Ice Pack to the Posterior Upper Neck. J Perianesth Nurs. 2022 Dec;37(6):774-777. doi: 10.1016/j.jopan.2021.12.010. Epub 2022 May 28. PMID 35637077
- [Background] Hymel N, Davies M. Evidence-Based Antiemetic Decision Tool for Management of Postoperative Nausea and Vomiting in Patients at High Risk of QT Prolongation and Patients Receiving Neurotransmitter-Modulating Medications. AANA J. 2020 Aug;88(4):312-318. PMID 32718430
- [Background] American Society of PeriAnesthesia Nurses PONV/PDNV Strategic Work Team. ASPAN'S evidence-based clinical practice guideline for the prevention and/or management of PONV/PDNV. J Perianesth Nurs. 2006 Aug;21(4):230-50. doi: 10.1016/j.jopan.2006.06.003. No abstract available. PMID 16935735
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162